CLINICAL TRIAL: NCT04551053
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the PI3Kδ Inhibitor Parsaclisib Plus Ruxolitinib in Participants With Myelofibrosis Who Have Suboptimal Response to Ruxolitinib
Brief Title: To Evaluate Efficacy and Safety of Parsaclisib and Ruxolitinib in Participants With Myelofibrosis Who Have Suboptimal Response to Ruxolitinib (LIMBER-304)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to futility.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB 50465-304/LIMBER-304; 2020-003415-98 (EudraCT Number); NCT04816565 (obsolete NCT alias)
Record Dates: First submitted 2020-09-11; First posted 2020-09-16 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Myelofibrosis; Primary Myelofibrosis; Post Essential Thrombocythemia Myelofibrosis; Post Polycythemia Vera Myelofibrosis
Keywords: INCB050465; ruxolitinib; parsaclisib; LIMBER; LIMBER-304; MF; MPN; Myeloproliferative Neoplasm; Myelofibrosis; Myoproliferative Neoplasms
MeSH Terms: conditions — Primary Myelofibrosis; Myeloproliferative Disorders | interventions — parsaclisib; ruxolitinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A : ruxolitinib +parsaclisib (Experimental): Participants will receive parsaclisib starting from Day 1 for the duration of study, while continuing to receive the stable dose of ruxolitinib they were taking for the 8 weeks prior to Day 1.
  Interventions: Drug: parsaclisib; Drug: ruxolitinib
- Group B : ruxolitinib + placebo (Placebo Comparator): Participants will receive placebo starting from Day 1 for the duration of study, while continuing to receive the stable dose of ruxolitinib they were taking for the 8 weeks prior to Day 1.
  Interventions: Drug: ruxolitinib; Drug: placebo

INTERVENTIONS:
Drug: parsaclisib — parsaclisib will be administered QD orally
  Other Names: INCB050465
  Arms: Group A : ruxolitinib +parsaclisib
Drug: ruxolitinib — ruxolitinib will be administered BID orally
  Other Names: Jakafi; Jakavi
Drug: placebo — placebo will be administered QD orally
  Arms: Group B : ruxolitinib + placebo

SUMMARY:
The purpose of the study is to compare the efficacy and safety of parsaclisib when combined with ruxolitinb versus placebo combined with ruxolitinib in participants with myelofibrosis who have suboptimal response while receiving ruxolitinib monotherapy.

DETAILED DESCRIPTION:
Prospective participants must be on stable doses of ruxolitinib ranging from 5 mg BID to 25 mg BID and will have been on that dose for at least the last 8 weeks prior to Day 1. At least 3 months duration of prior ruxolitinib is required. Participants must meet Protocol-defined criteria for suboptimal response to ruxolitinib monotherapy. After participants have been determined to be eligible for the study and completed the baseline symptom diary assessment for 7 days, they will be randomized to 1 of 2 treatment groups, with stratification for platelet count (≥ 100 × 10^9/L vs 50 to < 100 × 10^9/L inclusive) and DIPSS risk category (high vs intermediate-2 vs intermediate-1).

Once a participant has completed the week 24 assessments, the participant's treatment assignment will then be unblinded and if found to be placebo, the participant will have the opportunity to crossover to begin receiving parsaclisib, together with continued ruxolitinib, as long as hematology parameters are adequate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PMF, PPV-MF, or PET-MF.
* DIPSS risk category of intermediate-1, intermediate-2, or high.
* Treated with ruxolitinib for ≥ 3 months with a stable dose for at least the last 8 weeks prior to Day 1
* Palpable spleen of ≥ 5 cm below the left costal margin on physical examination at the screening visit.
* Active symptoms of MF at the screening visit, as demonstrated by the presence of a TSS of ≥ 10 using the Screening Symptom Form.
* Participants with an ECOG performance status score of 0, 1, or 2.
* Screening bone marrow biopsy specimen and pathology report(s) available that was obtained within the prior 2 months or willingness to undergo a bone marrow biopsy at screening/baseline; willingness to undergo bone marrow biopsy at Week 24 and every 24 weeks there after. Screening/baseline biopsy specimen must show diagnosis of MF.
* Life expectancy of at least 24 weeks.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Prior therapy with any drug that inhibits PI3K (examples of drugs targeting this pathway include but are not limited to INCB040093, idelalisib, duvelisib, buparlisib, copanlisib, and umbralisib).
* Use of experimental drug therapy for MF or any other standard drug used for MF (whether for treatment of MF or another indication) with the exception of ruxolitinib, within 3 months of starting study drug, and/or lack of recovery from all toxicities from previous therapy (except ruxolitinib) to Grade 1 or better.
* Inability to swallow food or any condition of the upper gastrointestinal tract that precludes administration of oral medications.
* Recent history of inadequate bone marrow reserve.
* Inadequate liver and renal function at screening.
* Active bacterial, fungal, parasitic, or viral infection that requires therapy.
* Active HBV or HCV infection that requires treatment or at risk for HBV reactivation.
* Known HIV infection.
* Uncontrolled, severe, or unstable cardiac disease that in the investigator's opinion may jeopardize the safety of the participant or compliance with the Protocol.
* Active invasive malignancy over the previous 2 years.
* Splenic irradiation within 6 months before receiving the first dose of study drug.
* Concurrent use of any prohibited medications.
* Active alcohol or drug addiction that would interfere with the ability to comply with the study requirements.
* Use of any potent CYP3A4 inhibitors or inducers within 14 days or 5 half lives(whichever is longer) before the first dose of study drug or anticipated during the study.
* Inadequate recovery from toxicity and/or complications from a major surgery before starting therapy.
* Currently breastfeeding or pregnant.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* History of Grade 3 or 4 irAEs from prior immunotherapy.
* Receipt of any live vaccine within 30 days of the first dose of study drug
* Unwillingness to receive RBC transfusions to treat low hemoglobin levels.
* Known hypersensitivity or severe reaction to parsaclisib or ruxolitinib or excipients of parsaclisib/matching placebo or ruxolitinib formulations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2024-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Assad, M.D., Study Director — Incyte Corporation
Locations (174):
- United States (35):
  - Sutter Health Alta Bates Summit Medical Center Absmc Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - CCARE, Fresno, California
  - California Research Institute (Cri), Los Angeles, California
  - Emad Ibrahim Md Inc, Redlands, California
  - Scripps Clinic, San Diego, California
  - Coastal Integrated Cancer Care - Cicc, San Luis Obispo, California
  - Stamford Hospital - Medical Oncology Hematology, Stamford, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Augusta University - Medical College of Georgia, Augusta, Georgia
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Kansas Hospital Authority, Westwood, Kansas
  - Tulane University, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Midamerica Cancer Care, Kansas City, Missouri
  - New Jersey Hematology Oncology Associates Llc, Brick, New Jersey
  - Morristown Medical Center - Atlantic Health System, Morristown, New Jersey
  - Westchester Medical Center Advanced Oncology, Hawthorne, New York
  - Mount Sinai School of Medicine, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Advent Health Hendersonville Park Ridge Hospital Hendersonville, Clyde, North Carolina
  - Duke Cancer Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Baptist Cancer Center, Memphis, Tennessee
  - Texas Oncology - Medical City Dallas, Dallas, Texas
  - Texas Oncology - Baylor Sammons Cancer Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Renovatio Clinical, Houston, Texas
  - Kelsey Seybold Clinic, Houston, Texas
  - Providence Regional Medical Center Everett, Everett, Washington
- Hanusch-Krankenhaus Wiener Gebietskrankenkasse, Vienna, Austria
- Belgium (4):
  - A.Z. St.-Jan A.V., Bruges
  - Jessa Ziekenhuis, Hasselt
  - AZ Delta, Roeselare
  - Chu Ucl Namur University Hospital Mont-Godinne, Yvoir
- China (29):
  - Peking University People'S Hospital (Pkuph) - Institute of Hematology, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - The First Peoples Hospital of Changzhou, Changzhou
  - Fujian Medical University Union Hospital, Fuzhou
  - Nanfang Hospital, Guangzhou
  - The First Affiliated Hospital of Zhejiang University, Hangzhou
  - Harbin Institute of Hematology and Oncology, Harbin
  - University of Science and Technology of China-First Affiliated Hospital (Anhui Provincial Hospital), Hefei
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot
  - Jinan Central Hospital, Jinan
  - The Second Affiliated Hospital of Kunming Medical University, Kunming
  - The First Hospital of Lanzhou University, Lanzhou
  - Lanzhou University Second Hospital, Lanzhou
  - Jiangxi Provincial of People Hospital, Nanchang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Jiangsu Province Hospital, Nanjing
  - The Affiliated Hospital of Qingdao University, Qingdao
  - The First Hospital of China Medical University, Shenyang
  - Shenzhen University Hospital, Shenzhen
  - Tianjin Medical University General Hospital, Tianjin
  - Institute of Hematology and Hospital of Blood Diseases, Chinese Academy of Medical Sciences and Pek, Tianjin
  - Union Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - Tongji Hospital Huazhong University of Science and Technology, Wuhan
  - The Second Affiliated Hospital of Xi an Jiaotong University, Xi'an
  - Yantai Yuhuangding Hospital, Yantai
  - Henan Provincial Peoples Hospital, Zhengzhou
  - Henan Cancer Hostipal, Zhengzhou
- Helsinki University Central Hospital, Helsinki, Finland
- France (10):
  - Centre Hospitalier Universitaire Grenoble Alpes (Chu Grenoble Alpes) - Hopital Albert Michallon, La Tronche
  - Chu de Limoges, Limoges
  - CHU Limoges - Hopital Duputren, Limoges
  - Centre Hospitalier Universitaire de Nantes (Chu de Nantes) - Hotel-Dieu, Nantes
  - Chu Nimes, Nîmes
  - Ap-Hp Groupe Hospitalier Saint-Louis Lariboisiere Fernand-Widal Site Saint Louis (Paris), Paris
  - Hospital Saint Antoine, Paris
  - Hospices Civils de Lyon Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut Universitaire Du Cancer de Toulouse Oncopole, Toulouse
  - Chu Vandoeuvre-Les-Nancy Hopital Brabois, Vandœuvre-lès-Nancy
- Germany (4):
  - Universitatsklinikum Bonn Aoer, Bonn
  - Universitaetsmedizin Greifswald, Greifswald
  - Universitatsklinikum Halle (Saale), Halle
  - Universitaetsmedizin Rostock, Rostock
- Hungary (3):
  - Semmelweis Egyetem, Budapest
  - Markhot Ferenc Korhaz, Eger
  - Petz Aladar County Teaching Hospital, Győr
- Israel (6):
  - Samson Assuta Ashdod University Hospital, Ashdod
  - Rambam Health Care Campus, Haifa
  - Hadassah Hebrew University Medical Center Ein Karem Hadassah, Jerusalem
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assuta Ramat Hahayal, Tel Aviv
- Italy (22):
  - Azienda Ospedaliera San Giuseppe Moscati, Avellino
  - Aou Policlinico Consorziale Di Bari, Bari
  - Lstituto Di Ematologia Lorenzo Ea.Seragnoli Universita Degli Studi Di Bologna - Policlinico S. Or, Bologna
  - Azienda Ospedaliera Di Rilievo Nazionale E Di Alta Specializzazione Garibaldi, Catania
  - University of Florence, Florence
  - Irccs Azienda Ospedaliera Universitaria San Martino, Genova
  - Fondazione Irccs Ca Granda Ospedale Maggiore, Milan
  - Universita Di Napoli Federico Ii, Napoli
  - Azienda Ospedaliero Universitaria Maggiore Della Carita Di Novara, Novara
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia - Cervello, Palermo
  - Ospedale S.Maria Della Misericordia, Perugia
  - Presidio Ospedaliero Pescara, Pescara
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Grande Ospedale Metropolitano Bianchi-Melacrino-Morelli, Reggio Calabria
  - Univ. Di Roma Facolta Di Armacia E Medicina, Roma
  - Policlinico Universitario Agostino Gemelli Universita Cattolica Del Sacro Cuore, Roma
  - Ospedale Sant. Eugenio, Roma
  - Policlinico Universitario Agostino Gemelli Universita Cattolica Del Sacro Cuore, Rome
  - Azienda Ospedaliera Universitaria Senese Policlinico Santa Maria Alle Scotte, Siena
  - Azienda Ospedaliera San Giuseppe Moscati, Taranto
  - Azienda Sanitaria Universitaria Friuli Centrale Asu Fc, Udine
  - A.O. Universitaria Ospedale Di Circolo E Fondazione Macchi, Varese
- Japan (18):
  - Kyushu University Hospital, Fukuoka
  - Japanese Red Cross Society Himeji Hospital, Himeji-shi
  - Kansai Medical University Hospital, Hirakata
  - Tokai University Hospital, Isehara
  - Juntendo University Hospital, Izunokuni
  - Kagoshima University Hospital, Kagoshima
  - Hospital of the University of Occupation and Environmental Health, Kitakyushu-shi
  - Kobe City Medical Center General Hospital, Kobe
  - Kumamoto Shinto General Hospital, Kumamoto
  - University of Miyazaki Hospital, Miyazaki
  - Japanese Red Cross Nagoya Daini Hospital, Nagoya
  - Osaka Metropolitan University Hospital, Osaka
  - Ogaki Municipal Hospital, Ōgaki
  - Dokkyo Medical University Saitama Medical Center, Saitama
  - Hokuyukai Sapporo Hokuyu Hospital, Sapporo
  - Juntendo University Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - University of Yamanashi Hospital, Yamanashi
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Akershus University Hospital, Lorenskog
- Poland (4):
  - Pratia Hematologia Katowice, Katowice
  - Samodzielny Publiczny Zoz Szpital Uniwersytecki W Krakowie, Krakow
  - Samodzielny Publiczny Szpital Kliniczny Nr 1, Lublin
  - Institute of Hematology and Transfusion Medicine, Warsaw
- Romania (2):
  - Spitalul Clinic Coltea - Clinica Hematologie, Bucharest
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Târgu Gânguleşti
- South Korea (4):
  - Pusan National University Yangsan Hospital, Busan
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St. Mary?S Hospital, Seoul
- Spain (15):
  - Hospital General Unviersitario de Alicante, Alicante
  - Ico Hospital Germans Trias I Pujol, Badalona
  - Hospital Del Mar, Barcelona
  - Hospital General Universitario Vall D Hebron, Barcelona
  - Institut Catala Doncologia Ico - Hospital Duran I Reynals Location, Barcelona
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Universitario 12 de Octubre, Madrid
  - Fundacion Jimenez Diaz University Hospital, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Virgen de La Arrixaca, Murcia
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitari I Politecnic La Fe, Valencia
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (3):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University (Ncku) Hospital, Tainan
- Turkey (Türkiye) (6):
  - Baskent University Adana Hospital, Adana
  - Gazi University Hospital Gazi University Faculty of Medicine, Ankara
  - Istanbul Medipol Universitesi Ibagcilar Medipol Mega Universitesi Hastanesi, Istanbul
  - Baskent University Istanbul Hospital, Istanbul
  - Ege University Hospital, Izmir
  - Ondokuz Mayis University Medicine Faculty, Samsun
- United Kingdom (5):
  - Grampian Health Board, Aberdeen
  - United Lincolnshire Hospitals, Boston
  - Gloucestershire Royal Hospital, Gloucester
  - University College London Hospitals Nhs Foundation Trust, London
  - James Cook University Hospital, Middlesbrough

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: Related Info — https://www.incyteclinicaltrials.com/limber/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted across sites in Austria, China, Finland, France, Germany, Hungary, Italy, Japan, South Korea, Norway, Poland, Spain, Turkey, the United Kingdom, and the United States.
Groups:
- Parsaclisib Plus Ruxolitinib: Participants were randomized to receive parsaclisib plus ruxolitinib beginning on Day 1. Participants received parsaclisib at a dose of 5 milligrams (mg) once daily (QD). Participants also received the stable dose of ruxolitinib they were taking for the 8 weeks prior to Day 1. Treatment with parsaclisib plus ruxolitinib continued for as long as the participant tolerated the regimen and did not meet any discontinuation criteria.
- Placebo Plus Ruxolitinib: Participants were randomized to receive placebo plus ruxolitinib beginning on Day 1 and continuing until Week 24. Participants received matching placebo at a dose of 5 mg QD and received the stable dose of ruxolitinib they were taking for the 8 weeks prior to Day 1. After 24 weeks, participants randomized to receive placebo plus ruxolitinib had to switch to treatment with parsaclisib plus ruxolitinib or discontinue treatment. Treatment continued for as long as the regimen was tolerated and the participant did not meet any discontinuation criteria. Participants who demonstrated worsening symptomatic splenomegaly could have switched to treatment with parsaclisib plus ruxolitinib early.
Period: Overall Study
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib
Started | 90 | 87
Completed | 0 | 0
Not Completed | 90 | 87
Not completed — Death | 10 | 9
Not completed — Lost to Follow-up | 0 | 2
Not completed — Study Terminated by Sponsor | 57 | 65
Not completed — Withdrawal by Subject | 12 | 5
Not completed — Adverse Event | 2 | 0
Not completed — Lack of Efficacy | 2 | 1
Not completed — Transitioned to Rollover per Protocol | 5 | 4
Not completed — Splenapendectomi | 1 | 0
Not completed — Medical Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib | Total
Number analyzed (Participants) | 90 | 87 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (9.88) | 62.3 (9.92) | 63.19 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 38 | 75
  Male | 53 | 49 | 102
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 45 | 52 | 97
  Black or African American | 1 | 1 | 2
  Asian | 37 | 26 | 63
  Not Reported | 7 | 8 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 10 | 12
  Not Hispanic or Latino | 70 | 57 | 127
  Not Reported | 7 | 4 | 11
  Unknown | 2 | 4 | 6
  Captured as "Other" in Database | 9 | 12 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving ≥25% Reduction in Spleen Volume From Baseline to Week 24 as Measured by Magnetic Resonance Imaging (MRI) (or Computed Tomography [CT] Scan in Applicable Participants)
Description: Participants had an MRI of the upper and lower abdomen and pelvis to determine the spleen volume. A CT scan was substituted for participants who were not candidates for MRI or when MRI was not readily available.
Time Frame: Baseline; Week 24
Population: Intent-to-Treat (ITT) Population: all randomized participants. Participants were analyzed if they had both Baseline and Week 24 measurements, or discontinued treatment before 03MAR2023 or switched treatment before Week 24, or reached Week 24 before 03MAR2023 but were missing Week 24 assessments. For participants who switched to parsaclisib plus ruxolitinib treatment early, data was truncated at the time of switch.
Measure: Number; unit: percentage of participants
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib
Number analyzed (Participants) | 72 | 72
percentage of participants | 16.7 | 9.7
Statistical Analysis 1: Comparison: Parsaclisib Plus Ruxolitinib vs Placebo Plus Ruxolitinib; Test type: Superiority — p-value for superiority is half of the CMH p-value; p = 0.2567, Cochran-Mantel-Haenszel — CMH test for un-equality stratified by Dynamic International Prognostic Scoring System (DIPSS) category (intermediate 1 versus intermediate 2 and high) and Baseline platelet count (≥100 × 10^9/Liters [L] versus 50 to <100 × 10^9/L inclusive); Odds Ratio (OR) = 1.80, 95% CI 2-sided [0.65 to 5.02]

2. Secondary Outcome: Percentage of Participants Who Have a ≥50% Reduction in Total Symptom Score (TSS) From Baseline to Week 24 as Measured by the Myelofibrosis Symptom Assessment Form v.4.0 (MFSAF v4.0) Diary
Description: Symptoms of myelofibrosis were assessed using the MFSAF v4.0 diary. The MFSAF v4.0 is composed of 7 individual symptom scores (fatigue, night sweats, itchiness, abdominal discomfort, pain under left ribs, early satiety, bone pain), each collected daily using a 0- (no symptoms) to 10-point (worst imaginable symptoms) scale. The daily TSS (0 to 70) is the sum of the 7 individual symptom scores collected in a day. A higher TSS corresponds to more severe symptoms. The TSS was marked as missing if there were any missing individual scores. Observations with missing dates were excluded from the analysis. The Baseline/Week 24 total score was defined as the average of the daily total scores from the last 7 days before the first dose of parsaclisib, placebo, or ruxolitinib/the Week 24 visit. The Baseline/Week 24 total score was marked as missing if there were ≥4 out of the 7 daily TSSs missing.
Time Frame: Baseline; Week 24
Population: ITT Population. Participants were analyzed if they had both Baseline and Week 24 measurements, or discontinued treatment before 03MAR2023 or switched treatment before Week 24, or reached Week 24 before 03MAR2023 but were missing Week 24 assessments. For participants who switched to parsaclisib plus ruxolitinib treatment early, data was truncated at the time of switch.
Measure: Number; unit: percentage of participants
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib
Number analyzed (Participants) | 70 | 71
percentage of participants | 17.1 | 14.1
Statistical Analysis 1: Comparison: Parsaclisib Plus Ruxolitinib vs Placebo Plus Ruxolitinib; Test type: Superiority — p-value for superiority is half of the CMH p-value; p = 0.5349, Cochran-Mantel-Haenszel — calculated from Cochran Mantel-Haenszel test for un-equality stratified by DIPSS category (intermediate 1 versus intermediate 2 and high) and Baseline platelet count (≥100 × 10^9/L versus 50 to <100 × 10^9/L inclusive); Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.53 to 3.39]

3. Secondary Outcome: Change in TSS From Baseline to Week 24 as Measured by the MFSAF v4.0 Diary
Description: Symptoms of myelofibrosis were assessed using the MFSAF v4.0 diary. The MFSAF v4.0 is composed of 7 individual symptom scores (fatigue, night sweats, itchiness, abdominal discomfort, pain under left ribs, early satiety, bone pain), each collected daily using a 0- (no symptoms) to 10-point (worst imaginable symptoms) scale. The daily TSS (0 to 70) is the sum of the 7 individual symptom scores collected in a day. A higher TSS corresponds to more severe symptoms. The TSS was marked as missing if there were any missing individual scores. Observations with missing dates were excluded from the analysis. The Baseline/Week 24 total score was defined as the average of the daily total scores from the last 7 days before the first dose of parsaclisib, placebo, or ruxolitinib/the Week 24 visit. The Baseline/Week 24 total score was marked as missing if there were ≥4 out of the 7 daily TSSs missing. Change from Baseline was calculated as the Week 24 value minus the Baseline value.
Time Frame: Baseline; Week 24
Population: ITT Population. Only participants with data available were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib
Number analyzed (Participants) | 88 | 82
scores on a scale
  Baseline | 17.2 (11.61) | 21.6 (14.28)
  Change from Baseline at Week 24: number analyzed (Participants) | 57 | 61
  Change from Baseline at Week 24 | -2.7 (8.67) | -2.7 (9.98)

4. Secondary Outcome: Time to the First ≥50% Reduction in TSS as Measured by the MFSAF v4.0 Diary
Description: Symptoms were assessed using the MFSAF v4.0 diary. The MFSAF v4.0 is composed of 7 individual symptom scores (fatigue, night sweats, itchiness, abdominal discomfort, pain under left ribs, early satiety, bone pain), each collected daily using a 0- (no symptoms) to 10-point (worst imaginable symptoms) scale. The daily TSS (0 to 70) is the sum of the 7 individual symptom scores collected in a day. A higher TSS corresponds to more severe symptoms. The TSS was marked as missing if there were any missing individual scores. Observations with missing dates were excluded from the analysis. The Baseline/Week 24 total score was defined as the average of the daily total scores from the last 7 days before the first dose of parsaclisib, placebo, or ruxolitinib/the Week 24 visit. The Baseline/Week 24 total scores was marked as missing if there were ≥4 out of the 7 daily TSSs missing. The 95% confidence interval was calculated using the Brookmeyer and Crowley's method with log-log transformation.
Time Frame: Baseline; up to Week 24
Population: ITT Population. For participants who switched to parsaclisib plus ruxolitinib treatment early, data was truncated at the time of switch. Participants with valid, calculated Baseline TSS and at least 1 postbaseline TSS who did not have a ≥50% reduction in TSS at the time of analysis were censored at the time of the last valid calculated TSS. If the participants had no valid, calculated Baseline or postbaseline TSS, they were censored at the date of randomization.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib
Number analyzed (Participants) | 90 | 87
days | NA [160.0 to NA] — The median and the upper limit of the confidence interval were not estimable because there were too few participants with a ≥50% reduction in TSS at the time of study termination. | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because there were too few participants with a ≥50% reduction in TSS at the time of study termination.
Statistical Analysis 1: Comparison: Parsaclisib Plus Ruxolitinib vs Placebo Plus Ruxolitinib; Test type: Superiority; p = 0.2224, Log Rank — calculated from log-rank test stratified by DIPSS category (intermediate 1 versus intermediate 2 and high) and Baseline platelet count (≥100 x 10^9/L versus 50 to <100 x 10^9/L inclusive)

5. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the interval between the randomization date and the date of death due to any cause.
Time Frame: up to 917 days
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib
Number analyzed (Participants) | 90 | 87
days | NA [NA to NA] — Due to study termination, the follow-up time was not long enough to estimate the median and the upper and lower limits of the confidence interval. | NA [NA to NA] — Due to study termination, the follow-up time was not long enough to estimate the median and the upper and lower limits of the confidence interval.

6. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug related. An AE could therefore be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A TEAE is defined as an AE reported for the first time or the worsening of a pre-existing event after the first dose of study treatment.
Time Frame: up to 917 days
Population: Safety Population: all randomized participants who received at least 1 dose of parsaclisib, placebo, or ruxolitinib. Treatment groups for this population were determined according to the actual treatment the participant received regardless of assigned study drug treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Swith to Parsaclisib: After 24 weeks, participants randomized to receive placebo plus ruxolitinib from Day 1 to Week 24 could have switched to treatment with parsaclisib plus ruxolitinib per the regimen received during the first 24 weeks of the study. Treatment continued for as long as the regimen was tolerated and the participant did not meet any discontinuation criteria. Participants who demonstrated worsening symptomatic splenomegaly could have switched to treatment with parsaclisb plus ruxolitinib early.
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib | Placebo Swith to Parsaclisib
Number analyzed (Participants) | 90 | 87 | 41
Participants | 81 | 76 | 33

7. Secondary Outcome: Number of Participants With Any Grade 3 or Higher TEAE
Description: An AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug related. A TEAE is defined as an AE reported for the first time or the worsening of a pre-existing event after the first dose of study treatment. The severity of AEs was assessed using Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Grades 1 through 5. Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2: moderate; minimal, local or noninvasive intervention indicated; limiting instrumental activities of daily living (ADL). Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4: life-threatening urgent intervention indicated. Grade 5: death related to AE.
Time Frame: up to 917 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib | Placebo Swith to Parsaclisib
Number analyzed (Participants) | 90 | 87 | 41
Participants | 54 | 37 | 18

8. Secondary Outcome: Time to the First ≥25% Reduction in Spleen Volume
Description: The time to the first ≥25% reduction in spleen volume is defined as the time from randomization to the first time participants had ≥25% reduction in spleen volume. Participants with a Baseline and post-Baseline MRI or CT scan who did not have ≥25% reduction in spleen volume at the time of analysis were censored at the time of the last MRI or CT scan. If the participants had no Baseline or post-Baseline MRI or CT scan, they were censored at the date of randomization.
Time Frame: up to 898 days
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib
Number analyzed (Participants) | 90 | 87
days | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants had a ≥25% reduction in spleen volume. | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants had a ≥25% reduction in spleen volume.

9. Secondary Outcome: Duration of Maintenance of a ≥25% Reduction in Spleen Volume
Description: The duration of ≥25% reduction from Baseline in spleen volume was defined as the interval between the first spleen volume measurement that was a ≥25% reduction from Baseline and the date of the first measurement that was no longer a ≥25% reduction from Baseline. If the end date was not observed before the database cutoff, the duration was censored at the last assessment.
Time Frame: up to 898 days
Population: ITT Population. Only those participants who had at least 1 measurement of ≥25% reduction from Baseline were to be analyzed. At the time of study termination, only a limited number of ≥25% reduction in spleen volume responses were observed; therefore, as specified in the Statistical Analysis Plan, analysis of duration of a 25% reduction in spleen volume was not performed.
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 917 days
Description: Treatment-emergent adverse events (TEAEs), defined as adverse events reported for the first time or the worsening of pre-existing events after the first dose of study treatment, have been reported for members of the Safety Population.
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib | Placebo Swith to Parsaclisib
All-Cause Mortality (participants affected / at risk) | 10/90 | 7/87 | 2/41
Serious Adverse Events (participants affected / at risk) | 33/90 | 15/87 | 8/41
Other Adverse Events (participants affected / at risk) | 71/90 | 58/87 | 25/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parsaclisib Plus Ruxolitinib (N=90) | Placebo Plus Ruxolitinib (N=87) | Placebo Swith to Parsaclisib (N=41)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 5 (5) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Necrotising colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 8 (11) | 2 (2) | 2 (2)
Pneumonia cytomegaloviral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia escherichia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Skin squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Subcapsular splenic haematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Transformation to acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ulcerative gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parsaclisib Plus Ruxolitinib (N=90) | Placebo Plus Ruxolitinib (N=87) | Placebo Swith to Parsaclisib (N=41)
Abdominal pain upper (Gastrointestinal disorders) | 8 (9) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 8 (9) | 3 (4) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 26 (38) | 20 (36) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 7 (8) | 4 (5) | 4 (5)
Asthenia (General disorders) | 7 (7) | 4 (4) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5) | 0 (0)
COVID-19 (Infections and infestations) | 16 (16) | 10 (10) | 6 (6)
Constipation (Gastrointestinal disorders) | 6 (7) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4) | 2 (2)
Cytomegalovirus infection (Infections and infestations) | 10 (10) | 0 (0) | 2 (2)
Cytomegalovirus test positive (Investigations) | 4 (4) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 9 (10) | 1 (4)
Dizziness (Nervous system disorders) | 7 (9) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (5) | 0 (0)
Fatigue (General disorders) | 5 (6) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 8 (8) | 4 (4) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 7 (7) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (8) | 7 (8) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 3 (3)
Neutrophil count decreased (Investigations) | 5 (7) | 3 (3) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 1 (1)
Platelet count decreased (Investigations) | 20 (33) | 14 (23) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 6 (10) | 0 (0)
Pyrexia (General disorders) | 13 (20) | 8 (14) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 6 (8) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (11) | 8 (10) | 8 (14)
White blood cell count decreased (Investigations) | 8 (12) | 7 (17) | 0 (0)

LIMITATIONS AND CAVEATS:
Following an interim analysis by an independent Data Monitoring Committee (DMC), the study was terminated early due to futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT04551053/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT04551053/SAP_002.pdf